CLINICAL TRIAL: NCT01709565
Title: Lactate Clearance and Mortality in Patients With Severe Sepsis and Septic Shock: Comparison by Hepatic Dysfunction
Brief Title: Lactate Clearance According to the Presence of Hepatic Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jo, Ik Joon, Associate Professor, Samsung Medical Center
Other Study IDs: SamsungMC
Record Dates: First submitted 2012-09-17; First posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Sepsis; Liver Failure
Keywords: Sepsis; Lactic acid; Shock; Resuscitation
MeSH Terms: conditions — Sepsis; Liver Failure; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Interleukin-1, Interleukin-6, Interleukin-10, TNF-alfa
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No hepatic dysfunction: No hepatic dysfunction, total plasma bilirubin ≤ 2.0 mg/dl
- Hepatic dysfunction: Hepatic dysfunction, total plasma bilirubin > 2.0 mg/dl

SUMMARY:
The purpose of this study is to compare lactate clearance in patients with severe sepsis and septic shock according to the presence of hepatic dysfunction.

DETAILED DESCRIPTION:
Lactate clearance is well known to be associated with mortality in patients with severe sepsis and septic shock. To normalize lactate levels is one of important goals of early resuscitation of sepsis patients.

Lactate clearance can be changed by various factors including patient characteristics, severity of shock, and treatment. In particular, hepatic dysfunction might impair the clearance of lactate because liver is a principal organ for lactate metabolism. However, an association between lactate clearance and hepatic failure has not been evaluated during initial resuscitation of patients with severe sepsis and septic shock. The primary goal of this study is to compare lactate clearance in patients with severe sepsis and septic shock according to the presence of hepatic dysfunction. The secondary goal is to evaluate if lactate clearance is associated with mortality even in patients with hepatic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented with septic shock or severe sepsis within 6 hours after emergency department arrival

Exclusion Criteria:

* Terminal malignancy or illness with a expected survival < 4 months
* Patients who previously signed "Do Not Resuscitate" or "Do Not Intubate" orders
* Patients who do not undergo the early goal-directed therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department and meeting criteria for severe sepsis or septic shock at Samsung Medical Center (a 1,960 bed, university-affiliated, tertiary referral hospital in Seoul, South Korea)
Sampling Method: Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Lactate clearance | at 6-hour from the time of enrollment
  [(initial lactate - delayed lactate)/ initial lactate] *100%

SECONDARY OUTCOMES:
In-hospital mortality | within the first 28-day after emergency department arrival

CONTACTS AND LOCATIONS:
Overall Officials: Ik Joon Jo, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Nguyen HB, Rivers EP, Knoblich BP, Jacobsen G, Muzzin A, Ressler JA, Tomlanovich MC. Early lactate clearance is associated with improved outcome in severe sepsis and septic shock. Crit Care Med. 2004 Aug;32(8):1637-42. doi: 10.1097/01.ccm.0000132904.35713.a7. PMID 15286537
- [Background] Levraut J, Ciebiera JP, Chave S, Rabary O, Jambou P, Carles M, Grimaud D. Mild hyperlactatemia in stable septic patients is due to impaired lactate clearance rather than overproduction. Am J Respir Crit Care Med. 1998 Apr;157(4 Pt 1):1021-6. doi: 10.1164/ajrccm.157.4.9705037. PMID 9563714
- [Background] De Jonghe B, Cheval C, Misset B, Timsit JF, Garrouste M, Montuclard L, Carlet J. Relationship between blood lactate and early hepatic dysfunction in acute circulatory failure. J Crit Care. 1999 Mar;14(1):7-11. doi: 10.1016/s0883-9441(99)90002-3. PMID 10102718
- [Background] Revelly JP, Tappy L, Martinez A, Bollmann M, Cayeux MC, Berger MM, Chiolero RL. Lactate and glucose metabolism in severe sepsis and cardiogenic shock. Crit Care Med. 2005 Oct;33(10):2235-40. doi: 10.1097/01.ccm.0000181525.99295.8f. PMID 16215376
- [Background] Kang YR, Um SW, Koh WJ, Suh GY, Chung MP, Kim H, Kwon OJ, Jeon K. Initial lactate level and mortality in septic shock patients with hepatic dysfunction. Anaesth Intensive Care. 2011 Sep;39(5):862-7. doi: 10.1177/0310057X1103900510. PMID 21970130
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Jones AE, Shapiro NI, Trzeciak S, Arnold RC, Claremont HA, Kline JA; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Lactate clearance vs central venous oxygen saturation as goals of early sepsis therapy: a randomized clinical trial. JAMA. 2010 Feb 24;303(8):739-46. doi: 10.1001/jama.2010.158. PMID 20179283